CLINICAL TRIAL: NCT05911841
Title: A Phase 2, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, 52 Week Study to Evaluate the Efficacy and Safety of LY3454738 in the Treatment of Adult Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Study of LY3454738 in the Treatment of Adult Participants With Moderate-to-Severe Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The decision to terminate the study was due to efficacy/effectiveness reasons.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18569; J4E-MC-FR01 (Other: Eli Lilly and Company); FR01 ISA (Other: Eli Lilly and Company); J4E-MC-IMMB Master Protocol (Other: Eli Lilly and Company); 2022-502888-38-00 (Other: EU Trial Number); NCT07020351 (obsolete NCT alias)
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo administered subcutaneously (SC) every two weeks (Q2W) from baseline to Week 14. Week 16 responders entered maintenance period and received placebo SC every four weeks (Q4W) until Week 40. Week 16 non-responders entered escape arm and received 800 milligrams (mg) of LY3454738 administered SC Q4W until Week 40.
  Interventions: Drug: LY3454738; Drug: Placebo
- 75 mg LY3454738 (Experimental): Participants received 75 mg of LY3454738 administered SC Q2W from baseline until Week 14. Week 16 responders entered maintenance period and received 150 mg of LY3454738 administered SC Q4W until Week 40. Week 16 non-responders entered escape arm and received 800 mg of LY3454738 administered SC Q4W until Week 40.
  Interventions: Drug: LY3454738
- 300 mg LY3454738 (Experimental): Participants received 300 mg of LY3454738 administered SC Q2W from baseline until Week 14. Week 16 responders entered maintenance period and continued receiving 300 mg of LY3454738 administered SC Q4W until Week 40. Week 16 non-responders entered escape arm and received 800 mg of LY3454738 administered SC Q4W until Week 40.
  Interventions: Drug: LY3454738
- 800 mg LY3454738 (Experimental): Participants received 800 mg of LY3454738 administered SC Q2W from baseline until Week 14. Week 16 responders entered maintenance period and were re-randomized to either receive 800 mg of LY3454738 or placebo administered SC Q4W until Week 40. Week 16 non-responders entered escape arm and received 800 mg of LY3454738 administered SC Q4W until Week 40.
  Interventions: Drug: LY3454738

INTERVENTIONS:
Drug: LY3454738 — Administered SC
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to describe the efficacy and safety of LY3454738 in adult participants with moderate-to-severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Are candidates for systemic therapy.

ISA specific:

* Have moderate-to-severe AD, defined as meeting all of the following criteria, at the first dosing visit:

  * EASI score greater than or equal to (≥)16
  * vIGA-AD score ≥3, and
  * ≥10% of BSA involvement (per EASI BSA).
* Have applied at least 1 emollient every day for at least 2 weeks before the day of the first dose of study intervention in this ISA and agree to daily use of at least 1 emollient continuously throughout the study.

Exclusion Criteria:

ISA specific:

* Have, in the screening period, any of the skin conditions, infections, or medical conditions listed under master IMMB.
* Are currently being treated with topical or systemic therapy
* Recent treatment with experimental (biologics and/or small molecules) - doesn't apply for subset of participants who must have been exposed to biologics and/or small molecules.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (66):
- United States (13):
  - Johnson Dermatology, Fort Smith, Arkansas
  - Arkansas Research Trials, North Little Rock, Arkansas
  - Dermatology Research Associates, Los Angeles, California
  - Encore Medical Research, Hollywood, Florida
  - Conquest Research, Winter Park, Florida
  - Allergy and Asthma Specialist, Owensboro, Kentucky
  - Revival Research Institute, LLC, Troy, Michigan
  - ActivMed Practices & Research, Inc., Portsmouth, New Hampshire
  - Metropolitan Dermatology - Clark, Kenilworth, New Jersey
  - Oregon Dermatology and Research Center, Portland, Oregon
  - DermDox Centers for Dermatology, Camp Hill, Pennsylvania
  - Progressive Clinical Research, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
- Canada (8):
  - Rejuvenation Dermatology, Calgary, Alberta
  - Rejuvenation Dermatology, Edmonton, Alberta
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - CCA Medical Research, Ajax, Ontario
  - Hamilton Allergy, Hamilton, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - FACET Dermatology, Toronto, Ontario
  - Alpha Recherche Clinique, Québec
- China (6):
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Renmin Hospital of Wuhan University, Wuhan
- Hungary (5):
  - Allergo-Derm Bakos Kft, Szolnok, Jász-Nagykun-Szolnok
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár, Somogy County
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely, Vas County
  - Medmare Bt, Veszprém, Veszprém City
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
- Japan (6):
  - Yasumoto Dermatology Clinic, Chikushino-shi, Fukuoka
  - Takagi Dermatological Clinic, Obihiro-shi, Hokkaido
  - Nomura Dermatology Clinic, Yokohama, Kanagawa
  - Dermatology and Ophthalmology Kume Clinic, Sakai, Osaka
  - Nihonbashi Sakura Clinic, Chuo-ku, Tokyo
  - Tachikawa Dermatology Clinic, Tachikawa, Tokyo
- Mexico (7):
  - Centro de Atención en Enfermedades Inflamatorias CATEI, Guadalajara, Jalisco
  - Cryptex Investigación Clínica S.A. de C.V., Cuauhtémoc, Ciudad de México, Mexico City
  - RM Pharma Specialists, Mexico City, Mexico City
  - Trials in Medicine, Mexico City, Mexico City
  - Eukarya PharmaSite, Monterrey, Nuevo León
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
- Poland (6):
  - Diamond Clinic, Krakow, Lesser Poland Voivodeship
  - MICS Centrum Medyczne Warszawa, Warsaw, Masovian Voivodeship
  - Specderm Poznanska, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - "DERMED" Centrum Medyczne Sp. z o.o., Lodz, Łódź Voivodeship
  - Dermoklinika - Centrum Medyczne spółka cywilna M. Kierstan, J. Narbutt, A. Lesiak, Lodz, Łódź Voivodeship
- South Korea (6):
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Bupyeong-gu, Incheon-gwangyeoksi [Incheon]
  - Korea University Ansan Hospital, Ansan-si, Kyǒnggi-do
  - Pusan National University Hospital, Busan, Pusan-Kwangyǒkshi
  - Chung-Ang University Hospital, Dongjak-gu, Seoul-teukbyeolsi [Seoul]
  - National Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Hallym University Kangnam Sacred Heart Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
- Taiwan (9):
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist, Kaohsiung
  - New Taipei Municipal TuCheng Hospital, New Taipei City, New Taipei
  - Chung Shan Medical University Hospital, Taichung, Taichung
  - Tri-Service General Hospital, Taipei City, Taipei
  - National Taiwan University Hospital - Hsinchu branch, Hsinchu
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of LY3454738 in the Treatment of Adult Participants With Moderate-to-Severe Atopic Dermatitis — https://trials.lilly.com/en-US/trial/407540

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Induction Period (16 weeks):
  Participants were randomly assigned to receive 75 mg or 300 mg or 800 mg of LY3454738 or placebo every 2 weeks (Q2W) subcutaneously (SC).
  Maintenance Period (28 weeks):
  At Week 16, participants who achieved a ≥50% improvement in EASI [EASI-50]) (responders) were reassigned as follows, continuing treatment through Week 40:
  • Responders from the 800 mg Q2W group were re-randomized to receive either 800 mg LY3454738 every 4 weeks (Q4W) or placebo Q4W.
  (continued)
Pre-assignment Details: * Responders from 300 mg Q2W arm received 300 mg LY3454738 Q4W.
  * Responders from 75 mg Q2W arm received 150 mg LY3454738 Q4W.
  * Responders from placebo Q2W arm received placebo Q4W.
  Escape Arm:
  Participants who didn't achieve EASI-50 at Week 16 (induction non-responders) or who didn't achieve ≥25% improvement from baseline in EASI at Week 20, 24, 28, 32, or 36 (maintenance non-responders) were assigned to Escape Arm. These participants received LY3454738 800 mg Q4W through Week 40.
Groups:
- Induction - Placebo Q2W: Induction Period: (Baseline - Week 16): Participants received SC injections of Placebo Q2W from Baseline until Week 14.
- Induction - LY3454738 75 mg Q2W: Induction Period (Baseline - Week 16): Participants received 75 mg of LY3454738 given SC Q2W from Baseline until Week 14.
- Induction - LY3454738 300 mg Q2W: Induction Period (Baseline - Week 16): Participants received 300 mg of LY3454738 given SC Q2W from Baseline until Week 14.
- Induction - LY3454738 800 mg Q2W: Induction Period (Baseline - Week 16): Participants received 800 mg of LY3454738 given SC Q2W from Baseline until Week 14.
- Maintenance Period - Placebo Q2W to Placebo Q4W: Maintenance Period (Week 16 - Week 44): Participants received Placebo administered SC Q4W from Week 16 to Week 40.
- Maintenance Period - LY3454738 75 mg Q2W to LY3454738 150 mg Q4W: Maintenance Period (Week 16 - Week 44): Participants received 150 mg LY3454738 SC Q4W from Week 16 to Week 40.
- Maintenance Period - LY3454738 300 mg Q2W to LY3454738 300 mg Q4W: Maintenance Period (Week 16 - Week 44): Participants received 300 mg LY3454738 SC Q4W from Week 16 to Week 40.
- Maintenance Period - LY3454738 800 mg Q2W to LY3454738 800 mg Q4W: Maintenance Period (Week 16 - Week 44): Participants received 800 mg LY3454738 SC Q4W from Week 16 to Week 40.
- Maintenance Period - LY3454738 800 mg Q2W to Placebo Q4W: Maintenance Period (Week 16 - Week 44): Participants received Placebo SC Q4W from Week 16 to Week 40.
- Escape Period - LY3454738 800 mg Q4W: Participants received 800 mg LY3454738 administered SC Q4W through Week 44.
Period: Induction Period
Arm/Group | Induction - Placebo Q2W | Induction - LY3454738 75 mg Q2W | Induction - LY3454738 300 mg Q2W | Induction - LY3454738 800 mg Q2W | Maintenance Period - Placebo Q2W to Placebo Q4W | Maintenance Period - LY3454738 75 mg Q2W to LY3454738 150 mg Q4W | Maintenance Period - LY3454738 300 mg Q2W to LY3454738 300 mg Q4W | Maintenance Period - LY3454738 800 mg Q2W to LY3454738 800 mg Q4W | Maintenance Period - LY3454738 800 mg Q2W to Placebo Q4W | Escape Period - LY3454738 800 mg Q4W
Started | 65 (Started includes Biologic- and small-molecule-naive n = 35; Biologic- and/or small-molecule-experienced n = 30.) | 31 (Started includes Biologic- and small-molecule-naive n = 30; Biologic- and/or small-molecule-experienced n = 1.) | 45 (Started includes Biologic- and small-molecule-naive n = 29; Biologic- and/or small-molecule-experienced n = 16.) | 93 (Started includes Biologic- and small-molecule-naive n = 60; Biologic- and/or small-molecule-experienced n = 33.) | 0 | 0 | 0 | 0 | 0 | 0
Received At Least One Dose of Study Drug | 65 | 31 | 45 | 93 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 53 (Completed includes Responders n = 22; Non responders n = 31.) | 26 (Completed includes Responders n = 13; Non responders n = 13.) | 21 (Completed includes Responders n = 8; Non responders n = 13.) | 76 (Completed includes Responders n = 39; Non responders n = 37.) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 12 | 5 | 24 | 17 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 2 | 0 | 14 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 3 | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Assigned Treatment by Mistake | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Period
Arm/Group | Induction - Placebo Q2W | Induction - LY3454738 75 mg Q2W | Induction - LY3454738 300 mg Q2W | Induction - LY3454738 800 mg Q2W | Maintenance Period - Placebo Q2W to Placebo Q4W | Maintenance Period - LY3454738 75 mg Q2W to LY3454738 150 mg Q4W | Maintenance Period - LY3454738 300 mg Q2W to LY3454738 300 mg Q4W | Maintenance Period - LY3454738 800 mg Q2W to LY3454738 800 mg Q4W | Maintenance Period - LY3454738 800 mg Q2W to Placebo Q4W | Escape Period - LY3454738 800 mg Q4W
Started | 0 (Participants were assigned to this arm only during Induction Period.) | 0 (Participants were assigned to this arm only during Induction Period.) | 0 (Participants were assigned to this arm only during Induction Period.) | 0 (Participants were assigned to this arm only during Induction Period.) | 22 (Only those participants who were responders in the Induction Period at Week 16 entered the Maintenance Period.) | 13 (Only those participants who were responders in the Induction Period at Week 16 entered the Maintenance Period.) | 8 (Only those participants who were responders in the Induction Period at Week 16 entered the Maintenance Period.) | 20 (Only those participants who were responders in the Induction Period at Week 16 entered the Maintenance Period.) | 19 (Only those participants who were responders in the Induction Period at Week 16 entered the Maintenance Period.) | 0
Received At Least One Dose of Study Drug | 0 | 0 | 0 | 0 | 22 | 13 | 8 | 20 | 19 | 0
Completed | 0 | 0 | 0 | 0 | 10 | 7 | 3 | 7 | 8 | 0
Not Completed | 0 | 0 | 0 | 0 | 12 | 6 | 5 | 13 | 11 | 0
Not completed — Enrolled to Escape Arm | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 4 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 11 | 5 | 1 | 7 | 7 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Escape Period
Arm/Group | Induction - Placebo Q2W | Induction - LY3454738 75 mg Q2W | Induction - LY3454738 300 mg Q2W | Induction - LY3454738 800 mg Q2W | Maintenance Period - Placebo Q2W to Placebo Q4W | Maintenance Period - LY3454738 75 mg Q2W to LY3454738 150 mg Q4W | Maintenance Period - LY3454738 300 mg Q2W to LY3454738 300 mg Q4W | Maintenance Period - LY3454738 800 mg Q2W to LY3454738 800 mg Q4W | Maintenance Period - LY3454738 800 mg Q2W to Placebo Q4W | Escape Period - LY3454738 800 mg Q4W
Started | 0 | 0 | 0 | 0 | 0 (Participants were assigned to this arm only during Maintenance Period.) | 0 (Participants were assigned to this arm only during Maintenance Period.) | 0 (Participants were assigned to this arm only during Maintenance Period.) | 0 (Participants were assigned to this arm only during Maintenance Period.) | 0 (Participants were assigned to this arm only during Maintenance Period.) | 105 (Only those participants who were non-responders in the Induction Period at Week 16 and who did not achieve at least 25% improvement in EASI at Week 20, 24, 28, 32, or 36 entered the Escape Period.)
Received At Least One Dose of Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 105
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 82
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Discontinued Due to Failure to Achieve an EASI-50 Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Site Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 34
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Induction - Placebo Q2W | Induction - LY3454738 75 mg Q2W | Induction - LY3454738 300 mg Q2W | Induction - LY3454738 800 mg Q2W | Total
Number analyzed (Participants) | 65 | 31 | 45 | 93 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (13.4) | 37.3 (12.4) | 36.1 (13.9) | 35.2 (12.6) | 36.4 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 13 | 21 | 39 | 101
  Male | 37 | 18 | 24 | 54 | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 2 | 12 | 28
  Not Hispanic or Latino | 57 | 24 | 40 | 80 | 201
  Unknown or Not Reported | 1 | 0 | 3 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 5 | 3 | 5 | 17
  Asian | 27 | 12 | 25 | 49 | 113
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 6 | 0 | 2 | 1 | 9
  White | 26 | 13 | 14 | 37 | 90
  More than one race | 1 | 1 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 5 | 3 | 6 | 9 | 23
  South Korea | 3 | 1 | 9 | 10 | 23
  Hungary | 3 | 3 | 0 | 5 | 11
  United States | 13 | 3 | 6 | 9 | 31
  China | 4 | 4 | 1 | 8 | 17
  Japan | 8 | 2 | 9 | 13 | 32
  Taiwan | 8 | 2 | 4 | 11 | 25
  Poland | 17 | 6 | 8 | 22 | 53
  Mexico | 4 | 7 | 2 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Biologic and Small Molecule Naive Participants Achieving Eczema Area and Severity Index (EASI) 75 (≥75% Reduction in EASI Score) at Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent, i.e., percentage of skin affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI-75 score was obtained by weight-averaging these 4 scores and will range from 0 (none) to 72 (severe).
  The EASI-75 responder is defined as a participant who achieves a ≥ 75% improvement from baseline in the EASI score.
Time Frame: Week 16
Population: All biologic and small-molecule-naive participants who were randomly assigned to study intervention and took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Induction - Placebo Q2W | Induction - LY3454738 75 mg Q2W | Induction - LY3454738 300 mg Q2W | Induction - LY3454738 800 mg Q2W
Number analyzed (Participants) | 35 | 30 | 29 | 60
Percentage of participants | 14.3 | 20.0 | 17.2 | 18.3

2. Secondary Outcome: Percentage of Biologic and Small Molecule Naive Participants Achieving EASI-50 (≥ 50% Reduction in EASI Score) at Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of AD - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  The EASI-50 responder is defined as a participant who achieves a ≥ 50% reduction from baseline in the EASI score.
Time Frame: Week 16
Population: All biologic and small-molecule-naive participants who were randomly assigned to study intervention and took at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Induction - Placebo Q2W | Induction - LY3454738 75 mg Q2W | Induction - LY3454738 300 mg Q2W | Induction - LY3454738 800 mg Q2W
Number analyzed (Participants) | 35 | 30 | 29 | 60
Percentage of participants | 28.6 | 40.0 | 24.1 | 45.0

3. Secondary Outcome: Percentage of Biologic and Small Molecule Naive Participants Achieving EASI-90 (≥ 90% Reduction in EASI Score) at Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of AD - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  The EASI-90 responder is defined as a participant who achieves a ≥ 90% reduction from baseline in the EASI score.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Induction - Placebo Q2W | Induction - LY3454738 75 mg Q2W | Induction - LY3454738 300 mg Q2W | Induction - LY3454738 800 mg Q2W
Number analyzed (Participants) | 35 | 30 | 29 | 60
Percentage of participants | 8.6 | 3.3 | 10.3 | 11.7

4. Secondary Outcome: Percentage of Biologic and Small Molecule Naive Participants Achieving SCORing Atopic Dermatitis (SCORAD) 75 at Week 16
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3)oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with a visual analogue scales (VAS) where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease.
  The SCORAD75 responder is defined as a participant who achieves a ≥ 75% improvement from baseline in the SCORAD score.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Induction - Placebo Q2W | Induction - LY3454738 75 mg Q2W | Induction - LY3454738 300 mg Q2W | Induction - LY3454738 800 mg Q2W
Number analyzed (Participants) | 35 | 30 | 29 | 60
Percentage of participants | 5.7 | 3.3 | 3.4 | 6.7

5. Secondary Outcome: Percentage of Biologic and Small Molecule Naive Participants Achieving SCORAD-90 at Week 16
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3)oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with a visual analogue scales (VAS) where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease.
  The SCORAD90 responder is defined as a participant who achieves a ≥ 90% improvement from baseline in the SCORAD score.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Induction - Placebo Q2W | Induction - LY3454738 75 mg Q2W | Induction - LY3454738 300 mg Q2W | Induction - LY3454738 800 mg Q2W
Number analyzed (Participants) | 35 | 30 | 29 | 60
Percentage of participants | 2.9 | 0.0 | 0.0 | 1.7

6. Secondary Outcome: Percentage of Biologic and Small Molecule Naive Participants Achieving Validated Investigator's Global Assessment for Atopic Dermatitis (vIGA-AD) of 0 or 1 at Week 16
Description: vIGA-AD is a standardized clinical tool used to measure the severity of AD. It is a static 5-point scale ranging from 0 to 4, used to grade overall disease severity. Higher viGA-AD scores represent more severe disease. The scale is as below:
  * 0-Clear: No inflammatory signs of atopic dermatitis (erythema, induration/papulation, lichenification, oozing/crusting). Post-inflammatory hyperpigmentation and/or hypopigmentation may be present.
  * 1-Almost Clear: Barely perceptible erythema, induration/papulation, and/or lichenification. No oozing/crusting.
  * 2-Mild: Slight but definite erythema (pink), induration/papulation, and/or lichenification. No oozing/crusting.
  * 3-Moderate: Clearly perceptible erythema (dull red), induration/papulation, and/or lichenification. Oozing and crusting may be present.
  * 4-Severe: Marked erythema (deep or bright red), induration/papulation, and/or lichenification. Disease is widespread in extent. Oozing or crusting may be present.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Induction - Placebo Q2W | Induction - LY3454738 75 mg Q2W | Induction - LY3454738 300 mg Q2W | Induction - LY3454738 800 mg Q2W
Number analyzed (Participants) | 35 | 30 | 29 | 60
Percentage of participants | 8.6 | 6.7 | 6.9 | 15.0

7. Secondary Outcome: Percentage of Biologic and Small Molecule Naive Participants Achieving ≥4-point Improvement From Baseline in Itch Numeric Rating Scale (NRS) in the Subset of Biologic and Small Molecule Naive Participants With ≥4-point Itch NRS at Baseline
Description: Percentage of biologic and small molecule naive participants achieving ≥4-point improvement from baseline in Itch NRS in the Subset of biologic and small molecule naive participants with ≥4-point Itch NRS at Baseline were reported.
  The Itch NRS is a an 11-point scale used by participants to rate their worst itch severity over the past 24 hours with 0 indicating "No itch" and 10 indicating "Worst itch imaginable."
Time Frame: Baseline, Week 16
Population: All biologic and small-molecule-naive participants who were randomly assigned to study intervention and took at least one dose of study drug in the subset of participants with ≥4-point Itch NRS at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Induction - Placebo Q2W | Induction - LY3454738 75 mg Q2W | Induction - LY3454738 300 mg Q2W | Induction - LY3454738 800 mg Q2W
Number analyzed (Participants) | 31 | 25 | 19 | 44
Percentage of participants | 12.9 | 24.0 | 5.3 | 6.8

8. Secondary Outcome: Mean Percent Change From Baseline in EASI in Biologic and Small Molecule Naive Participants
Description: Mean percent change from baseline in EASI in biologic and small molecule naive participants was reported.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Induction - Placebo Q2W | Induction - LY3454738 75 mg Q2W | Induction - LY3454738 300 mg Q2W | Induction - LY3454738 800 mg Q2W
Number analyzed (Participants) | 35 | 30 | 29 | 60
Percent change | -25.2 (7.10) | -37.2 (6.39) | -25.3 (6.83) | -40.1 (4.76)
Statistical Analysis 1: Comparison: Induction - Placebo Q2W vs Induction - LY3454738 75 mg Q2W; Test type: Superiority; Mean Difference (Final Values) = -12.0, 95% CI 2-sided [-30.6 to 6.6]
Statistical Analysis 2: Comparison: Induction - Placebo Q2W vs Induction - LY3454738 300 mg Q2W; Test type: Superiority; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-19.4 to 19.2]
Statistical Analysis 3: Comparison: Induction - Placebo Q2W vs Induction - LY3454738 800 mg Q2W; Test type: Superiority; Mean Difference (Final Values) = -14.9, 95% CI 2-sided [-31.6 to 1.7]

9. Secondary Outcome: Mean Percent Change From Baseline in SCORAD in Biologic and Small Molecule Naive Participants
Description: Mean percent change from baseline in SCORAD in biologic and small molecule naive participants was reported.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Induction - Placebo Q2W | Induction - LY3454738 75 mg Q2W | Induction - LY3454738 300 mg Q2W | Induction - LY3454738 800 mg Q2W
Number analyzed (Participants) | 35 | 30 | 29 | 60
Percent change | -16.6 (4.86) | -21.0 (4.65) | -15.2 (5.01) | -26.6 (3.58)
Statistical Analysis 1: Comparison: Induction - Placebo Q2W vs Induction - LY3454738 75 mg Q2W; Test type: Superiority; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-17.6 to 8.7]
Statistical Analysis 2: Comparison: Induction - Placebo Q2W vs Induction - LY3454738 300 mg Q2W; Test type: Superiority; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-12.3 to 15.1]
Statistical Analysis 3: Comparison: Induction - Placebo Q2W vs Induction - LY3454738 800 mg Q2W; Test type: Superiority; Mean Difference (Final Values) = -9.9, 95% CI 2-sided [-21.8 to 1.9]

10. Secondary Outcome: Percentage of Biologic and Small Molecule Experienced Participants Achieving EASI-75 at Week 16
Description: as for outcome 1
Time Frame: Week 16
Population: All biologic and small-molecule-experienced participants who were randomly assigned to study intervention and took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Induction - Placebo Q2W | Induction - LY3454738 75 mg Q2W | Induction - LY3454738 300 mg Q2W | Induction - LY3454738 800 mg Q2W
Number analyzed (Participants) | 30 | 1 | 16 | 33
Percentage of participants | 20.0 | 0.0 | 6.2 | 12.1

11. Secondary Outcome: Pharmacokinetics (PK): Serum Trough Concentrations of LY3454738 at Week 16
Description: PK: Serum trough concentrations of LY3454738 were reported.
Time Frame: Day 113 post Day 1 Dose
Population: All biologic and/or small molecule experienced or biologic-and-small-molecule naïve participants who were randomly assigned to study intervention and took at least 1 dose of LY3454738 and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (μg/mL)
Groups:
- LY3454738 75 mg: All participants who received 75 mg of LY3454738 given SC Q2W were included in this arm.
- LY3454738 300 mg: All participants who received 300 mg of LY3454738 given SC Q2W were included in this arm.
- LY3454738 800 mg: All participants who received 800 mg of LY3454738 given SC Q2W were included in this arm.
Arm/Group | LY3454738 75 mg | LY3454738 300 mg | LY3454738 800 mg
Number analyzed (Participants) | 26 | 22 | 77
micrograms per milliliter (μg/mL) | 12.1 (7.01) | 56.2 (18.5) | 151 (56.2)

ADVERSE EVENTS:
Time Frame: Baseline Through Follow-up (Up To 52 Weeks)
Description: All randomized participants. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | Induction - Placebo Q2W | Induction - LY3454738 75 mg Q2W | Induction - LY3454738 300 mg Q2W | Induction - LY3454738 800 mg Q2W | Maintenance Period - Placebo Q2W to Placebo Q4W | Maintenance Period - LY3454738 75 mg Q2W to LY3454738 150 mg Q4W | Maintenance Period - LY3454738 300 mg Q2W to LY3454738 300 mg Q4W | Maintenance Period - LY3454738 800 mg Q2W to LY3454738 800 mg Q4W | Maintenance Period - LY3454738 800 mg Q2W to Placebo Q4W | Escape Period - LY3454738 800 mg Q4W
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/31 | 0/45 | 0/93 | 0/22 | 0/13 | 0/8 | 0/20 | 0/19 | 0/105
Serious Adverse Events (participants affected / at risk) | 3/65 | 1/31 | 1/45 | 1/93 | 1/22 | 1/13 | 0/8 | 1/20 | 0/19 | 0
Other Adverse Events (participants affected / at risk) | 35/65 | 19/31 | 20/45 | 52/93 | 13/22 | 7/13 | 4/8 | 7/20 | 6/19 | 39/105
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Induction - Placebo Q2W | Induction - LY3454738 75 mg Q2W | Induction - LY3454738 300 mg Q2W | Induction - LY3454738 800 mg Q2W | Maintenance Period - Placebo Q2W to Placebo Q4W | Maintenance Period - LY3454738 75 mg Q2W to LY3454738 150 mg Q4W | Maintenance Period - LY3454738 300 mg Q2W to LY3454738 300 mg Q4W | Maintenance Period - LY3454738 800 mg Q2W to LY3454738 800 mg Q4W | Maintenance Period - LY3454738 800 mg Q2W to Placebo Q4W | Escape Period - LY3454738 800 mg Q4W
Anaphylactic shock (Immune system disorders) | 0/65 (0) | 1/31 (1) | 0/45 (0) | 0/93 (0) | 0/22 (0) | 0/13 (0) | 0/8 (0) | 0/20 (0) | 0/19 (0) | 0/105 (0)
Pneumonia (Infections and infestations) | 0/65 (0) | 0/31 (0) | 0/45 (0) | 0/93 (0) | 0/22 (0) | 0/13 (0) | 0/8 (0) | 1/20 (1) | 0/19 (0) | 0/105 (0)
Traumatic pain (Injury, poisoning and procedural complications) | 0/65 (0) | 0/31 (0) | 1/45 (1) | 0/93 (0) | 0/22 (0) | 0/13 (0) | 0/8 (0) | 0/20 (0) | 0/19 (0) | 0/105 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0/65 (0) | 0/31 (0) | 0/45 (0) | 0/93 (0) | 1/22 (1) | 0/13 (0) | 0/8 (0) | 0/20 (0) | 0/19 (0) | 0/105 (0)
Device dislocation (Product Issues) | 1/65 (1) | 0/31 (0) | 0/45 (0) | 0/93 (0) | 0/22 (0) | 0/13 (0) | 0/8 (0) | 0/20 (0) | 0/19 (0) | 0/105 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0/65 (0) | 0/31 (0) | 0/45 (0) | 1/93 (1) | 0/22 (0) | 0/13 (0) | 0/8 (0) | 0/20 (0) | 0/19 (0) | 0/105 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0/65 (0) | 0/31 (0) | 0/45 (0) | 0/93 (0) | 0/22 (0) | 1/13 (1) | 0/8 (0) | 0/20 (0) | 0/19 (0) | 0/105 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1/65 (1) | 0/31 (0) | 0/45 (0) | 0/93 (0) | 0/22 (0) | 0/13 (0) | 0/8 (0) | 0/20 (0) | 0/19 (0) | 0/105 (0)
Hypotension (Vascular disorders) | 1/65 (1) | 0/31 (0) | 0/45 (0) | 0/93 (0) | 0/22 (0) | 0/13 (0) | 0/8 (0) | 0/20 (0) | 0/19 (0) | 0/105 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Induction - Placebo Q2W (N=65) | Induction - LY3454738 75 mg Q2W (N=31) | Induction - LY3454738 300 mg Q2W (N=45) | Induction - LY3454738 800 mg Q2W (N=93) | Maintenance Period - Placebo Q2W to Placebo Q4W (N=22) | Maintenance Period - LY3454738 75 mg Q2W to LY3454738 150 mg Q4W (N=13) | Maintenance Period - LY3454738 300 mg Q2W to LY3454738 300 mg Q4W (N=8) | Maintenance Period - LY3454738 800 mg Q2W to LY3454738 800 mg Q4W (N=20) | Maintenance Period - LY3454738 800 mg Q2W to Placebo Q4W (N=19) | Escape Period - LY3454738 800 mg Q4W (N=105)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lens dislocation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Administration site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Administration site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Administration site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Condition aggravated (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (11) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 4 (6)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to animal (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atopy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Milk allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vulvovaginitis (Infections and infestations) | 0/28 (0) | 0/13 (0) | 0/21 (0) | 0/39 (0) | 0/11 (0) | 1/7 (1) | 0/5 (0) | 0/10 (0) | 0/6 (0) | 0/38 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis infected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Fungal foot infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 4 (4) | 3 (4) | 10 (10) | 3 (4) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 4 (5)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Puncture site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 2 (2) | 0 (0) | 7 (9) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 4 (4)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0/28 (0) | 0/13 (0) | 0/21 (0) | 1/39 (2) | 0/11 (0) | 0/7 (0) | 0/5 (0) | 0/10 (0) | 0/6 (0) | 0/38 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Barotitis media (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid scar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural erythema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagogastroscopy (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/28 (0) | 0/13 (0) | 0/21 (0) | 0/39 (0) | 0/11 (0) | 0/7 (0) | 0/5 (0) | 1/10 (1) | 0/6 (0) | 0/38 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (8) | 2 (2) | 2 (3) | 6 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0/28 (0) | 0/13 (0) | 0/21 (0) | 0/39 (0) | 0/11 (0) | 0/7 (0) | 0/5 (0) | 0/10 (0) | 0/6 (0) | 1/38 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/28 (0) | 0/13 (0) | 0/21 (0) | 2/39 (2) | 0/11 (0) | 0/7 (0) | 0/5 (0) | 1/10 (2) | 0/6 (0) | 0/38 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary calcification (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Androgenetic alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail deformation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intra-uterine contraceptive device removal (Surgical and medical procedures) | 0/28 (0) | 0/13 (0) | 0/21 (0) | 0/39 (0) | 0/11 (0) | 0/7 (0) | 0/5 (0) | 0/10 (0) | 0/6 (0) | 1/38 (1)
Tooth extraction (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (4):
  • Study Protocol: IMMB(b) Protocol (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT05911841/Prot_000.pdf
  • Study Protocol: FR01(c) Protocol (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT05911841/Prot_001.pdf
  • Statistical Analysis Plan: FR01 Statistical Analysis Plan (Version 3) (2025-05-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT05911841/SAP_002.pdf
  • Statistical Analysis Plan: IMMB Statistical Analysis Plan (Version 1) (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT05911841/SAP_003.pdf